CLINICAL TRIAL: NCT03625895
Title: Agrylin Capsules 0.5 mg Drug Use-Result Survey
Brief Title: Agrylin Drug Use-Result Survey
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: SHP422-406
Record Dates: First submitted 2018-08-08; First posted 2018-08-10 (Actual); Results first posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2022-05

CONDITIONS: Essential Thrombocythemia (ET)
MeSH Terms: conditions — Thrombocythemia, Essential

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anagrelide hydrochloride: Participants who received treatment with Anagrelide hydrochloride will be evaluated for this study. Participants will receive interventions as part of routine medical care.

SUMMARY:
The objective of this survey is to collect data to evaluate the safety and efficacy of anagrelide hydrochloride in the post-marketing phase in participants diagnosed with Essential Thrombocythemia (ET).

DETAILED DESCRIPTION:
Anagrelide hydrochloride Drug Use-Result Survey

ELIGIBILITY:
Inclusion Criteria:

- All cases who received treatment with Agrylin.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with essential thrombocythemia (ET) being treated with agrylin will be evaluated for this study.
Sampling Method: Non-Probability Sample
Enrollment: 1826 (Actual)
Dates: Start 2014-11-25 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (300):
- Japan (300):
  - Gamagori-city, Gamagōri, Aichi-ken
  - Handa City, Handa, Aichi-ken
  - Hekinan-city, Hekinan, Aichi-ken
  - Ichinomiya-city, Ichinomiya, Aichi-ken
  - Komaki-city, Komaki, Aichi-ken
  - Nagakute-city, Nagakute, Aichi-ken
  - Nagoya-city, Nagoya, Aichi-ken
  - Nishio-city, Nishio, Aichi-ken
  - Okazaki-city, Okazaki, Aichi-ken
  - Obu-city, Ōbu, Aichi-ken
  - Seto-city, Seto, Aichi-ken
  - Toyoake-city, Toyoake, Aichi-ken
  - Toyohashi-city, Toyohashi, Aichi-ken
  - Toyota-city, Toyota, Aichi-ken
  - Akita-city, Akita, Akita
  - Noshiro-city, Noshiro, Akita
  - Yurihonjo-city, Yurihonjō, Akita
  - Aomori-city, Aomori, Aomori
  - Hachinohe-city, Hachinohe, Aomori
  - Asahi-city, Asahi, Chiba
  - Chiba-city, Chiba, Chiba
  - Funabashi-city, Funabashi, Chiba
  - Ichihara-city, Ichihara, Chiba
  - Ichikawa-city, Ichikawa, Chiba
  - Inzai-city, Inzai, Chiba
  - Kamogawa-city, Kamogawa, Chiba
  - Kashiwa-city, Kashiwa, Chiba
  - Kisarazu-city, Kisarazu, Chiba
  - Matsudo-city, Matsudo, Chiba
  - Narita-city, Narita, Chiba
  - Oamishirasato-city, Ōamishirasato, Chiba
  - Sakura-city, Sakura, Chiba
  - Urayasu-city, Urayasu, Chiba
  - Matsuyama-city, Matsuyama, Ehime
  - Toon-city, Tōon, Ehime
  - Fukui-city, Fukui-shi, Fukui
  - Obama-city, Obama, Fukui
  - Tsuruga-city, Tsuruga, Fukui
  - Asakura-gun, Asakura-gun, Fukuoka
  - Fukuoka-city, Fukuoka, Fukuoka
  - Iizuka-city, Iizuka, Fukuoka
  - Kasuga-city, Kasuga, Fukuoka
  - Kitakyushu-city, Kitakyushu, Fukuoka
  - Koga-city, Koga, Fukuoka
  - Kurume-city, Kurume, Fukuoka
  - Munakata-city, Munakata, Fukuoka
  - Date-city, Date, Fukushima
  - Fukushima-city, Fukushima, Fukushima
  - Minamisoma-city, Minamisoma-city, Fukushima
  - Soma-city, Sōma, Fukushima
  - Gifu-city, Gifu, Gifu
  - Gujo-city, Gujō, Gifu
  - Kani-city, Kani, Gifu
  - Minokamo-city, Minokamo, Gifu
  - Ogaki-city, Ōgaki, Gifu
  - Seki-city, Sekimachi, Gifu
  - Tajimi-city, Tajimi, Gifu
  - Takayama-city, Takayama, Gifu
  - Annaka-city, Annaka, Gunma
  - Fujioka-city, Fujioka, Gunma
  - Maebashi-city, Maebashi, Gunma
  - Ota-city, Ōta, Gunma
  - Tomioka-city, Tomioka, Gunma
  - Fukuyama-city, Fukuyama, Hiroshima
  - Higashihiroshima-city, Higashihiroshima, Hiroshima
  - Hiroshima-city, Hiroshima, Hiroshima
  - Kure-city, Kure, Hiroshima
  - Mihara-city, Mihara, Hiroshima
  - Otake-city, Ōtake, Hiroshima
  - Sera-gun, Sera-gun, Hiroshima
  - Asahikawa-city, Asahikawa, Hokkaido
  - Chitose-city, Chitose, Hokkaido
  - Furano-city, Furano, Hokkaido
  - Hakodate-city, Hakodate, Hokkaido
  - Kushiro-city, Kushiro, Hokkaido
  - Muroran-city, Muroran, Hokkaido
  - Nemuro-city, Nemuro, Hokkaido
  - Obihiro-city, Obihiro, Hokkaido
  - Otaru-city, Otaru, Hokkaido
  - Sapporo-city, Sapporo, Hokkaido
  - Tomakomai-city, Tomakomai, Hokkaido
  - Wakkanai-city, Wakkanai, Hokkaido
  - Akashi-city, Akashi, Hyōgo
  - Ako-city, Ako, Hyōgo
  - Amagasaki-city, Amagasaki, Hyōgo
  - Himeji-city, Himeji, Hyōgo
  - Itami-city, Itami, Hyōgo
  - Kasai-city, Kasai, Hyōgo
  - Kobe-city, Kobe, Hyōgo
  - Nishinomiya-city, Nishinomiya, Hyōgo
  - Nishiwaki-city, Nishiwaki, Hyōgo
  - Sasayama-city, Sasayama, Hyōgo
  - Sumoto-city, Sumoto, Hyōgo
  - Takarazuka-city, Takarazuka, Hyōgo
  - Tamba-city, Tamba, Hyōgo
  - Tanba-city, Tanba, Hyōgo
  - Higashiibaraki-gun, Higashiibaraki-gun, Ibaraki
  - Hitachi-city, Hitachi, Ibaraki
  - Hitachinaka-city, Hitachi-Naka, Ibaraki
  - Inashiki-gun, Inashiki-gun, Ibaraki
  - Ishioka-city, Ishioka, Ibaraki
  - Kasama-city, Kasama, Ibaraki
  - Koga-city, Koga, Ibaraki
  - Mito-city, Mito, Ibaraki
  - Moriya-city, Moriya, Ibaraki
  - Namegata-city, Namegata, Ibaraki
  - Toride-city, Toride, Ibaraki
  - Tsuchiura-city, Tsuchiura, Ibaraki
  - Tsukuba-city, Tsukuba, Ibaraki
  - Ushiku-city, Ushiku, Ibaraki
  - Kahoku-gun, Kahoku-gun, Ishikawa-ken
  - Kanazawa-city, Kanazawa, Ishikawa-ken
  - Komatsu-city, Komatsu, Ishikawa-ken
  - Nanao-city, Nanao, Ishikawa-ken
  - Kitakami-city, Kitakami, Iwate
  - Morioka-city, Morioka, Iwate
  - Ninohe-city, Ninohe, Iwate
  - Oshu-city, Ōshū, Iwate
  - Kanonji-city, Kan’onjichō, Kagawa-ken
  - Sakaide-city, Sakaidechō, Kagawa-ken
  - Sanuki-city, Sanuki, Kagawa-ken
  - Takamatsu-city, Takamatsu, Kagawa-ken
  - Kagoshima-city, Kagoshima, Kagoshima-ken
  - Minamisatsuma-city, Minamisatsuma, Kagoshima-ken
  - Oshima-gun, Oshima-gun, Kagoshima-ken
  - Chigasaki-city, Chigasaki, Kanagawa
  - Ebina-city, Ebina, Kanagawa
  - Fujisawa-city, Fujisawa, Kanagawa
  - Isehara-city, Isehara, Kanagawa
  - Kamakura-city, Kamakura, Kanagawa
  - Kawasaki-city, Kawasaki, Kanagawa
  - Sagamihara-city, Sagamihara, Kanagawa
  - Yokohama-city, Yokohama, Kanagawa
  - Yokosuka-city, Yokosuka, Kanagawa
  - Aki-city, Aki, Kochi
  - Kochi-city, Kochi, Kochi
  - Nankoku-city, Nankoku, Kochi
  - Shimanto-city, Shimanto, Kochi
  - Tosa-city, Tosa, Kochi
  - Amakusa-city, Amakusa, Kumamoto
  - Arao-city, Arao, Kumamoto
  - Kumamoto-city, Kumamoto, Kumamoto
  - Fukuchiyama-city, Fukuchiyama, Kyoto
  - Kyoto-city, Kyoto, Kyoto
  - Maizuru-city, Maizuru, Kyoto
  - Uji-city, Uji, Kyoto
  - Yawata-city, Yawata, Kyoto
  - Ise-city, Ise, Mie-ken
  - Kumano-city, Kumano, Mie-ken
  - Kuwana-city, Kuwana, Mie-ken
  - Matsusaka-city, Matsusaka, Mie-ken
  - Suzuka-city, Suzuka, Mie-ken
  - Tsu-city, Tsu, Mie-ken
  - Yokkaichi-city, Yokkaichi, Mie-ken
  - Natori-city, Natori-shi, Miyagi
  - Osaki-city, Ōsaki, Miyagi
  - Sendai-city, Sendai, Miyagi
  - Miyakonojo-city, Miyakonojō, Miyazaki
  - Miyazaki-city, Miyazaki, Miyazaki
  - Kitaazumi-gun, Kitaazumi-gun, Nagano
  - Matsumoto-city, Matsumoto, Nagano
  - Nagano-city, Nagano, Nagano
  - Saku-city, Saku, Nagano
  - Suwa-city, Suwa, Nagano
  - Suzaka-city, Suzaka, Nagano
  - Iki-city, Iki, Nagasaki
  - Isahaya-city, Isahaya, Nagasaki
  - Nagasaki-city, Nagasaki, Nagasaki
  - Omura-city, Ōmura, Nagasaki
  - Sasebo-city, Sasebo, Nagasaki
  - Ikoma-city, Ikoma, Nara
  - Nara-city, Nara, Nara
  - Sakurai-city, Sakurai, Nara
  - Tenri-city, Tenri, Nara
  - Yamatokoriyama-city, Yamatokōriyama, Nara
  - Itoigawa-city, Itoigawa, Niigata
  - Joetsu-city, Jōetsu, Niigata
  - Kashiwazaki-city, Kashiwazaki, Niigata
  - Minamiuonuma-city, Minamiuonuma, Niigata
  - Nagaoka-city, Nagaoka, Niigata
  - Niigata-city, Niigata, Niigata
  - Ojiya-city, Ojiya, Niigata
  - Sado-city, Sado, Niigata
  - Shibata-city, Shibata, Niigata
  - Tsubame-city, Tsubame, Niigata
  - Bungotakada-city, BungoTakada, Oita Prefecture
  - Nakatsu-city, Nakatsu, Oita Prefecture
  - Oita-city, Ōita, Oita Prefecture
  - Kurashiki-city, Kurashiki, Okayama-ken
  - Maniwa-city, Maniwa, Okayama-ken
  - Okayama-city, Okayama, Okayama-ken
  - Tamano-city, Tamano, Okayama-ken
  - Kunigami-gun, Kunigami-gun, Okinawa
  - Nago-city, Nago, Okinawa
  - Naha-city, Naha, Okinawa
  - Nakagami-gun, Nakagami-gun, Okinawa
  - Okinawa-city, Okinawa, Okinawa
  - Uruma-city, Uruma, Okinawa
  - Higashiosaka-city, Higashiosaka, Osaka
  - Hirakata-city, Hirakata, Osaka
  - Ikeda-city, Ikeda, Osaka
  - Izumiootsu-city, Izumiootsu-city, Osaka
  - Izumiotsu-city, Izumiōtsu, Osaka
  - Izumisano-city, Izumisano, Osaka
  - Kaizuka-city, Kaizuka, Osaka
  - Kawachinagano-city, Kawachi-Nagano, Osaka
  - Kishiwada-city, Kishiwada, Osaka
  - Mino-city, Mino-city, Osaka
  - Moriguchi-city, Moriguchi, Osaka
  - Neyagawa-city, Neyagawa, Osaka
  - Osaka-city, Osaka, Osaka
  - Sakai-city, Sakai, Osaka
  - Osakasayama-city, Sayama, Osaka
  - Suit-city, Suit-city, Osaka
  - Suita-city, Suita, Osaka
  - Takatsuki-city, Takatsuki, Osaka
  - Tondabayashi-city, Tondabayashi, Osaka
  - Toyonaka-city, Toyonaka, Osaka
  - Saga-city, Saga, Saga-ken
  - Chichibu-city, Chichibu, Saitama
  - Fukaya-city, Fukaya, Saitama
  - Hasuda-city, Hasuda, Saitama
  - Iruma-gun, Iruma-gun, Saitama
  - Kawagoe-city, Kawagoe, Saitama
  - Kawaguchi-city, Kawaguchi, Saitama
  - Kitaadachi-gun, Kitaadachi-gun, Saitama
  - Koshigaya-city, Koshigaya, Saitama
  - Niiza-city, Niiza, Saitama
  - Soka-city, Sōka, Saitama
  - Tokorozawa-city, Tokorozawa, Saitama
  - Tsurugashima-city, Tsurugashima, Saitama
  - Moriyama-city, Moriyama, Shiga
  - Nagahama-city, Nagahama, Shiga
  - Omihachiman-city, Ōmihachiman, Shiga
  - Otsu-city, Ōtsu, Shiga
  - Ritto-city, Rittō, Shiga
  - Gotsu-city, Gōtsuchō, Shimane
  - Hamada-city, Hamada, Shimane
  - Izumo-city, Izumo, Shimane
  - Masuda-city, Masuda, Shimane
  - Matsue-city, Matsue, Shimane
  - Nita-gun, Nita-gun, Shimane
  - Unnan-city, Unnan, Shimane
  - Fujieda-city, Fujieda, Shizuoka
  - Hamamatsu-city, Hamamatsu, Shizuoka
  - Iwata-city, Iwata, Shizuoka
  - Izunokuni-city, Izunokuni, Shizuoka
  - Mishima-city, Mishima, Shizuoka
  - Shizuoka-city, Shizuoka, Shizuoka
  - Ashikaga-city, Ashikaga, Tochigi
  - Sano-city, Sano, Tochigi
  - Shimotsuga-gun, Shimotsuga-gun, Tochigi
  - Shimotsuke-city, Shimotsuke, Tochigi
  - Utsunomiya-city, Utsunomiya, Tochigi
  - Yaita-city, Yaita, Tochigi
  - Itano-gun, Itano-gun, Tokushima
  - Naruto-city, Narutochō-mitsuishi, Tokushima
  - Tokushima-city, Tokushima, Tokushima
  - Adachi-ku, Adachi-ku, Tokyo
  - Akishima-city, Akishima, Tokyo
  - Bunkyo-ku, Bunkyo-ku, Tokyo
  - Chiyoda-ku, Chiyoda-ku, Tokyo
  - Chofu-city, Chōfu, Tokyo
  - Chuo-ku, Chuo-ku, Tokyo
  - Edogawa-ku, Edogawa-ku, Tokyo
  - Fuchu-city, Fuchū, Tokyo
  - Hachioji-city, Hachiōji, Tokyo
  - Itabashi-ku, Itabashi-ku, Tokyo
  - Katsushika-ku, Katsushika-ku, Tokyo
  - Koganei-city, Koganei, Tokyo
  - Meguro-ku, Meguro-ku, Tokyo
  - Minato-ku, Minato-ku, Tokyo
  - Nerima-ku, Nerima-ku, Tokyo
  - Ome-city, Ōme, Tokyo
  - Setagaya-ku, Setagaya-ku, Tokyo
  - Shibuya-ku, Shibuya-ku, Tokyo
  - Shinagawa-ku, Shinagawa-ku, Tokyo
  - Shinjuku-ku, Shinjuku-ku, Tokyo
  - Sumida-ku, Sumida-ku, Tokyo
  - Tachikawa-city, Tachikawa, Tokyo
  - Taito-ku, Taito-ku, Tokyo
  - Tottori-city, Tottori-shi, Tottori
  - Kurobe-city, Kurobe-shi, Toyama
  - Oyabe-city, Oyabe, Toyama
  - Takaoka-city, Takaoka, Toyama
  - Tonami-city, Tonami, Toyama
  - Toyama-city, Toyama, Toyama
  - Arida-gun, Arida-gun, Wakayama
  - Gobo-city, Gobō, Wakayama
  - Higashimuro-gun, Higashimuro-gun, Wakayama
  - Nishimuro-gun, Nishimuro-gun, Wakayama
  - Tanabe-city, Tanabe, Wakayama
  - Wakayama-city, Wakayama, Wakayama
  - Yamagata-city, Yamagata, Yamagata
  - Hofu-city, Hōfu, Yamaguchi
  - Oshima-gun, Oshima-gun, Yamaguchi
  - Shimonoseki-city, Shimonoseki, Yamaguchi
  - Shunan-city, Shūnan, Yamaguchi
  - Yamaguchi-city, Yamaguchi, Yamaguchi
  - Kofu-city, Kofu, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fd24db2bf003ab46ad8?idFilter=%5B%22SHP422-406%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant s took part in the survey at 513 investigative sites in Japan, from 25 November 2014 to 11 March 2021.
Pre-assignment Details: Participants with a historical diagnosis of essential thrombocythemia were enrolled. Participants received anagrelide hydrochloride as part of a routine medical care.
Period: Overall Study
Arm/Group | Anagrelide Hydrochloride
Started | 1826
Completed | 1241
Not Completed | 585
Not completed — Protocol Violation | 585

BASELINE CHARACTERISTICS:
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 1241
Age, Customized [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    ≤ 17 | 7
    18 - 64 | 443
    ≥ 65 | 790
    Unknown | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 705
  Male | 536
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Japan | 1241
History of Essential Thrombocythemia [Mean (Standard Deviation); unit: years] | 5.7 (6.10)
Platelet Count at Registration [Mean (Standard Deviation); unit: 10^4 platelets/µL] | 97.7 (45.63)
Janus kinase (JAK)-2 Status [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    Positive | 374
    Negative | 276
    Not Done | 584
    Unknown | 7
Prior Thrombocythemia Therapy [Count of Participants; unit: Participants]
  Had No Prior Thrombocythemia Therapy (Treatment Naïve) | 242
  Had Prior Thrombocythemia Therapy | 999
Pregnancy Test at Baseline [Count of Participants; unit: Participants] — Unknown: Data could not be collected. Population: The number analyzed is the number of participants with data available for analysis.
  Participants
    number analyzed (Participants) | 705
    Positive | 0
    Negative | 4
    Not Done/Unknown | 701
Medical History/Complication [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history or complications were classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history or complications included all medical history or complications except for those mentioned above.
  Participants
    Had No Medical History/Complication | 445
    Had Medical History/Complication | 796

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had One or More Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Time Frame: From start of study drug administration up to 12 months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 1241
Participants | 776

2. Primary Outcome: Number of Participants Who Had One or More Serious Adverse Event
Description: A serious AE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria.
Time Frame: From start of study drug administration up to 12 months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 1241
Participants | 234

3. Primary Outcome: Number of Participants Who Had One or More Adverse Drug Reactions
Description: AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. Adverse drug reaction refers to AE related to administered drug.
Time Frame: From start of study drug administration up to 12 months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 1241
Participants | 628

4. Primary Outcome: Number of Participants Who Had One or More Serious Adverse Drug Reactions
Description: A serious AE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria. Serious adverse drug reaction refers to serious AE that are related to administered drug.
Time Frame: From start of study drug administration up to 12 months
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 1241
Participants | 100

5. Primary Outcome: Percentage of Participants Who Responded in Platelet Count
Description: Percentage of participants who responded in platelet count was assessed. A response was defined as platelet counts to <60 x10^4 platelet/mcrL beyond 3 months after the start of study drug administration.
Time Frame: From 3 months after the start of study drug administration, up to 12 months
Population: Efficacy assessment population, The efficacy assessment population was defined as participants who completed the survey and had efficacy data at baseline and post-baseline time points available.
Measure: Number; unit: Percentage of Participants
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 880
Percentage of Participants | 61.02

6. Primary Outcome: Percentage of Participants With Normalization in Platelet Count
Description: Percentage of participants with normalization in platelet count was assessed. Normalization was defined as platelet counts to <40 x10^4 platelets/mcrL beyond 3 months after the start of study drug administration.
Time Frame: From 3 months after the start of study drug administration, up to 12 months
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 1039
Percentage of Participants | 28.97

7. Secondary Outcome: Percentage of Participants With at Least 50% Reduction in Platelet Count
Description: Participants who achieved at least 50% reduction in platelet count from their baseline during the 1-year observation period was assessed.
Time Frame: From start of study drug administration up to 12 months
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Anagrelide Hydrochloride
Number analyzed (Participants) | 1203
Percentage of Participants | 38.90

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 12 months
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Anagrelide Hydrochloride
All-Cause Mortality (participants affected / at risk) | 47/1241
Serious Adverse Events (participants affected / at risk) | 234/1241
Other Adverse Events (participants affected / at risk) | 477/1241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anagrelide Hydrochloride (N=1241)
Anaemia (Blood and lymphatic system disorders) | 4
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 3
Acute coronary syndrome (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 6
Angina pectoris (Cardiac disorders) | 8
Angina unstable (Cardiac disorders) | 3
Aortic valve incompetence (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 6
Bradycardia (Cardiac disorders) | 1
Bundle branch block bilateral (Cardiac disorders) | 1
Cardiac aneurysm (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 19
Cardiac failure acute (Cardiac disorders) | 3
Cardiac failure chronic (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 11
Cardiac failure high output (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 5
Myocardial ischaemia (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 3
Right ventricular failure (Cardiac disorders) | 1
Stress cardiomyopathy (Cardiac disorders) | 3
Torsade de pointes (Cardiac disorders) | 1
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Autoimmune thyroiditis (Endocrine disorders) | 1
Basedow's disease (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Angle closure glaucoma (Eye disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 3
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Peritoneal haematoma (Gastrointestinal disorders) | 1
Rectal ulcer (Gastrointestinal disorders) | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Condition aggravated (General disorders) | 1
Death (General disorders) | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Oedema (General disorders) | 1
Pyrexia (General disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholangitis acute (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Liver disorder (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Hepatitis E (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 3
Pseudomembranous colitis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Septic shock (Infections and infestations) | 1
Vascular device infection (Infections and infestations) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 2
Tendon rupture (Injury, poisoning and procedural complications) | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 6
Electrocardiogram T wave inversion (Investigations) | 1
Pancreatic enzymes increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 6
Marasmus (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered state of consciousness (Nervous system disorders) | 1
Brain stem infarction (Nervous system disorders) | 1
Cerebral artery stenosis (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 6
Cerebral infarction (Nervous system disorders) | 17
Cerebrovascular stenosis (Nervous system disorders) | 1
Dementia Alzheimer's type (Nervous system disorders) | 1
Dementia with Lewy bodies (Nervous system disorders) | 2
Encephalopathy (Nervous system disorders) | 1
Lacunar infarction (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1
Putamen haemorrhage (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Thrombotic cerebral infarction (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 5
Bipolar I disorder (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Renal disorder (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 7
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 13
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 7
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 4
Dialysis (Surgical and medical procedures) | 1
Aortic dissection (Vascular disorders) | 2
Aortic thrombosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Extremity necrosis (Vascular disorders) | 2
Haematoma (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Internal haemorrhage (Vascular disorders) | 1
Polyarteritis nodosa (Vascular disorders) | 1
Prinzmetal angina (Vascular disorders) | 3
Raynaud's phenomenon (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anagrelide Hydrochloride (N=1241)
Headache (Nervous system disorders) | 180
Palpitations (Cardiac disorders) | 154
Anaemia (Blood and lymphatic system disorders) | 76
Diarrhoea (Gastrointestinal disorders) | 67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT03625895/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT03625895/SAP_001.pdf